CLINICAL TRIAL: NCT01857804
Title: Surgical Treatment of Peri-implantitis With and Without Adjunctive Use of Antibiotics : a Controlled and Randomized Clinical Study
Brief Title: Surgical Treatment of Peri-implantitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: olivier1
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; surgical therapy; systemic antibiotics; local antiseptics
MeSH Terms: conditions — Peri-Implantitis | interventions — Amoxicillin; chlorhexidine gluconate; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- antibiotics and local antiseptics (Experimental): systemic antibiotics (2 x 750mg amoxicillin/day) + implant surface decontamination with chlorhexidine gluconate 0,2%
  Interventions: Drug: Amoxicillin; Drug: Chlorhexidine gluconate
- antibiotics without local antiseptics (Experimental): systemic antibiotics (2 x 750mg amoxicillin/day) + implant surface decontamination with saline
  Interventions: Drug: Amoxicillin
- local antiseptics no antibiotics (Experimental): no systemic antibiotics + implant surface decontamination with chlorhexidine gluconate 0,2%
  Interventions: Drug: Chlorhexidine gluconate
- no antibiotics and no local antiseptics (Placebo Comparator): no systemic antibiotics + implant surface decontamination with saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Amoxicillin — In the test group a systemic antibiotic regimen will be initiated at 3 days before surgery and continued for 10 days. (2 x 750mg amoxicillin/day or 2 x 1g amoxicillin/day depending on the weight of the patient)
  Other Names: systemic antibiotics
  Arms: antibiotics and local antiseptics; antibiotics without local antiseptics
Drug: Chlorhexidine gluconate — The exposed implant surfaces will be cleaned 3 minutes with antiseptics (chlorhexidine gluconate 0,2%) during the surgical treatment
  Other Names: chlorhexidine gluconate 0,2%
  Arms: antibiotics and local antiseptics; local antiseptics no antibiotics
Drug: Saline — The exposed implant surfaces will be cleaned 3 minutes with saline during the surgical treatment
  Arms: no antibiotics and no local antiseptics

SUMMARY:
The objective of this randomized controlled clinical trial is to evaluate the outcome of treatment of peri-implantitis with or without systemic antibiotics.

Specific aims are to analyze (i) the effect of systemic antibiotics and local antiseptics on the healing process, and (ii) the risk for recurrence of disease following surgical treatment of peri-implantitis.

DETAILED DESCRIPTION:
The study is designed as a randomized controlled clinical trial. 100 patients with severe peri-implantitis at one or more implants needing surgical treatment will be recruited. All individuals have to show unremarkable general health and not been using any antibiotics during the 6 months preceding the current examination.

The patients will be randomly assigned to the following :

* test group (T) : surgical treatment with systemic antibiotics,
* control group (C) : surgical treatment without systemic antibiotics. A stratification protocol will be applied regarding distribution of smokers. Two subgroups will be formed among test and control subjects.
* saline group (T1 and C1) : the exposed implant surfaces will be cleaned 3 minutes with saline during the surgical treatment, and,
* antiseptics group (T2 and C2) : the exposed implant surfaces will be cleaned 3 minutes with antiseptics (chlorhexidine 0,2%) during the surgical treatment.

A stratification protocol will be applied regarding distribution of smokers.

Following the baseline examination, patients will randomly be assigned to the various treatment group. Samples from the subgingival microbiota will be obtained before surgical therapy.

All patients will be enrolled in a hygiene program including professional supragingival implant/tooth cleaning using rubber cups and polishing paste and oral hygiene instructions.

The following clinical parameters will be measured at baseline using a periodontal probe: plaque index, Bleeding on Probing, probing depth measured from the mucosal margin to the bottom of the probable pocket and mucosal recession measured from a fixed landmark on the implant to the mucosal margin.

The measurements will be made at 4 aspects of each implant. In the test group (T) a systemic antibiotic regimen will be initiated at 3 days before surgery and continued for 10 days. (2 x 750mg amoxicillin/day or 2 x 1g amoxicillin/day depending on the weight of the patient) Intra-oral radiographs will be taken at 2 weeks and 1 year after surgical therapy.

The professional implant/tooth cleaning and reinforcement of oral hygiene will be performed at 2 weeks, 1, 2, 3, 6, and 12 months after treatment.

Examination of clinical outcome variables will be performed at 3, 6 and 12 months after surgical therapy. Microbiological samples will be obtained at the same time points. Radiographs are taken 2 weeks post surgical and at the one year examination.

Primary outcomes variables include: (i) clinical signs of resolution of peri-implantitis (pocket closure and absence of BoP), (ii) recurrence of the disease (BoP and increase in PPD) and (iii) further loss in marginal bone support, and (iiii) microbiological findings.

ELIGIBILITY:
Inclusion Criteria:

* peri-implant probing pocket depth > 7 mm on at least one aspect of the implant, together with BOP and/or suppuration,
* marginal bone loss > 3mm as detected in radiographs.

Exclusion Criteria:

* implant mobility,
* peri-implantitis associated bone defects not suitable for pocket elimination therapy,
* systemic diseases that could influence the outcome of the therapy,
* penicillin allergy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
pocket closure | 6 months, 1 year
  absence of probing pocket depth > 5 mm and no bleeding on probing
bone level stability | 1 year
  no further peri-implant marginal bone loss in the observation period.

SECONDARY OUTCOMES:
Quantitative and qualitative change in levels of the peri-implant microflora | 3 months, 6 months, 1 year
  Quantitative and qualitative change in levels of the peri-implant microflora

CONTACTS AND LOCATIONS:
Overall Officials: Tord Berglundh, Professor, Study Chair — Department of Periodontology, Institute of Odontology, The sahlgrenska academy, University of Gothenburg
Locations (1):
- Department of Periodontology, Institute of Odontology, Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Background] Albouy JP, Abrahamsson I, Persson LG, Berglundh T. Implant surface characteristics influence the outcome of treatment of peri-implantitis: an experimental study in dogs. J Clin Periodontol. 2011 Jan;38(1):58-64. doi: 10.1111/j.1600-051X.2010.01631.x. Epub 2010 Nov 24. PMID 21092053
- [Background] Ericsson I, Persson LG, Berglundh T, Edlund T, Lindhe J. The effect of antimicrobial therapy on periimplantitis lesions. An experimental study in the dog. Clin Oral Implants Res. 1996 Dec;7(4):320-8. doi: 10.1034/j.1600-0501.1996.070404.x. PMID 9151598
- [Background] Gualini F, Berglundh T. Immunohistochemical characteristics of inflammatory lesions at implants. J Clin Periodontol. 2003 Jan;30(1):14-8. doi: 10.1034/j.1600-051x.2003.300103.x. PMID 12702106
- [Background] Leonhardt A, Dahlen G, Renvert S. Five-year clinical, microbiological, and radiological outcome following treatment of peri-implantitis in man. J Periodontol. 2003 Oct;74(10):1415-22. doi: 10.1902/jop.2003.74.10.1415. PMID 14653386
- [Background] Mombelli A, Feloutzis A, Bragger U, Lang NP. Treatment of peri-implantitis by local delivery of tetracycline. Clinical, microbiological and radiological results. Clin Oral Implants Res. 2001 Aug;12(4):287-94. doi: 10.1034/j.1600-0501.2001.012004287.x. English, French, German. PMID 11488856
- [Background] Mombelli A, Lang NP. Antimicrobial treatment of peri-implant infections. Clin Oral Implants Res. 1992 Dec;3(4):162-8. doi: 10.1034/j.1600-0501.1992.030402.x. PMID 1298430
- [Background] Persson LG, Ericsson I, Berglundh T, Lindhe J. Guided bone regeneration in the treatment of periimplantitis. Clin Oral Implants Res. 1996 Dec;7(4):366-72. doi: 10.1034/j.1600-0501.1996.070410.x. PMID 9151604
- [Background] Persson LG, Ericsson I, Berglundh T, Lindhe J. Osseintegration following treatment of peri-implantitis and replacement of implant components. An experimental study in the dog. J Clin Periodontol. 2001 Mar;28(3):258-63. doi: 10.1034/j.1600-051x.2001.028003258.x. PMID 11284540
- [Background] Persson LG, Mouhyi J, Berglundh T, Sennerby L, Lindhe J. Carbon dioxide laser and hydrogen peroxide conditioning in the treatment of periimplantitis: an experimental study in the dog. Clin Implant Dent Relat Res. 2004;6(4):230-8. doi: 10.1111/j.1708-8208.2004.tb00039.x. PMID 15841583
- [Background] Wetzel AC, Vlassis J, Caffesse RG, Hammerle CH, Lang NP. Attempts to obtain re-osseointegration following experimental peri-implantitis in dogs. Clin Oral Implants Res. 1999 Apr;10(2):111-9. doi: 10.1034/j.1600-0501.1999.100205.x. PMID 10219130
- [Derived] Adly MS, Adly AS, Rasheed AM, Adly AS. CAN COMBINING LOW LEVEL LASER THERAPY WITH COMPUTER GUIDED FLAPLESS PIEZOSURGICAL OSTEOTOMY ACHIEVE A PAINLESS IMPLANT SURGERY? FINDINGS OF SPLIT MOUTH RANDOMIZED CONTROLLED TRIAL. J Evid Based Dent Pract. 2022 Sep;22(3):101730. doi: 10.1016/j.jebdp.2022.101730. Epub 2022 Apr 18. PMID 36162887
- [Derived] Graziani F, Cei S, Orlandi M, Gennai S, Gabriele M, Filice N, Nisi M, D'Aiuto F. Acute-phase response following full-mouth versus quadrant non-surgical periodontal treatment: A randomized clinical trial. J Clin Periodontol. 2015 Sep;42(9):843-852. doi: 10.1111/jcpe.12451. Epub 2015 Oct 1. PMID 26309133
- [Derived] Carcuac O, Derks J, Charalampakis G, Abrahamsson I, Wennstrom J, Berglundh T. Adjunctive Systemic and Local Antimicrobial Therapy in the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial. J Dent Res. 2016 Jan;95(1):50-7. doi: 10.1177/0022034515601961. Epub 2015 Aug 18. PMID 26285807